CLINICAL TRIAL: NCT03239119
Title: A Phase 3, Randomized, Double-Blind,Placebo-Controlled, Multicenter Study to Examine the Effect on Glucose Control (HbA1c) and Safety of rE-4 in Subjects With Type 2 Diabetes Mellitus Treated With Metformin, a Sulfonylurea, or Metformin and Sulfonylurea Combination
Brief Title: The Effectivity and Safety Study of rExenatide-4 in Chinese Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rE-4201706/PRO
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Type2 Diabetes Mellitus
Keywords: rE-4; Exenatide; Metformin; Sulfonylurea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rE-4 5 mcg (Experimental): Placebo, then rE-4 5 mcg, then rE-4 5 mcg
  Interventions: Biological: rE-4 5 mcg
- rE-4 10 mcg (Experimental): Placebo, then rE-4 5 mcg, then rE-4 10 mcg
  Interventions: Biological: rE-4 10 mcg
- Placebo 5 mcg (Placebo Comparator): Placebo 5 mcg, then Placebo 5 mcg, then Placebo 5 mcg
  Interventions: Biological: Placebo 5 mcg
- Placebo 10 mcg (Placebo Comparator): Placebo 5 mcg, then Placebo 5 mcg, then Placebo 10 mcg
  Interventions: Biological: Placebo 10 mcg

INTERVENTIONS:
Biological: rE-4 5 mcg — Placebo Lead In (5 mcg) for 4 weeks / rE-4 5 mcg for 4 weeks / rE-4 5 mcg for 26 weeks - All are subcutaneously injected twice daily
  Other Names: rExenatide-4
  Arms: rE-4 5 mcg
Biological: rE-4 10 mcg — Placebo Lead In (5 mcg) for 4 weeks / rE-4 5 mcg for 4 weeks / rE-4 10 mcg for 26 weeks - All are subcutaneously injected twice daily
  Other Names: rExenatide-4
  Arms: rE-4 10 mcg
Biological: Placebo 5 mcg — Placebo Lead In (5 mcg) for 4 weeks / Placebo 5 mcg for 4 weeks / Placebo 5 mcg for 26 weeks - All are subcutaneously injected twice daily
  Arms: Placebo 5 mcg
Biological: Placebo 10 mcg — Placebo Lead In (5 mcg) for 4 weeks / Placebo 5 mcg for 4 weeks / Placebo 10 mcg for 26 weeks - All are subcutaneously injected twice daily
  Arms: Placebo 10 mcg

SUMMARY:
This research is a randomized, double-blind,controlled trial. 456 Chinese subjects with Type 2 Diabetes Mellitus will be enrolled in the trial.

DETAILED DESCRIPTION:
This is a multicenter, randomized, blinded, placebo-controlled study to assess the effects on glucose control of rE-4 as compared to placebo in patients with type 2 diabetes. Patients will be randomized into one of two rE-4 treatment arms or to placebo treatment and will continue with their required existing diabetes medications (metformin, a sulfonylurea or metformin and a sulfonylurea combination) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. T2DM
2. 7.0% ≤ HbA1c ≤ 11.0% at screening
3. FPG ≤13.8 mmol/L
4. 19 kg/m2 < BMI <35.0 kg/m2 at screening
5. All subjects provided written informed consent before participation

Exclusion Criteria:

1. T1DM
2. Patients treated previously with Exenatide or GLP-1 similar
3. At screening visit alanine aminotransferase (ALT) or alkaline phosphatase (AST) more than 2.5 ULN
4. At screening visit estimated glomerular filtration rate (eGFR) ≤ 60 mL/min or Triglyceride(TG)≥ 5 mmol/L
5. Pancreatitis, cholecystitis, gallstones and other gastrointestinal diseases
6. Within the last 12 months prior to screening visit: history of stroke, myocardial infarction, unstable angina, or heart failure requiring hospitalization. Planned coronary, carotid or peripheral artery revascularisation procedures to be performed during the study period
7. History of digestive diseases (e.g.pancreatitis, cholecystitis or gallstones)
8. Patients with severe renal impairment or end-stage renal disease
9. Uncontrolled or inadequately controlled hypertension (systolic blood pressure above 180 mmHg or diastolic blood pressure above 110 mmHg) at screening visit.
10. Use of weight loss drugs within 3 months prior to screening visit
11. Have been treated with exogenous insulin, α-glucosidase, corticosteroid, DPP-4 inhibitor or pramlintide acetate within the 3 months prior to screening.
12. Severe gastrointestinal disease (e.g., gastroparesis)
13. Pregnancy or lactation, women of childbearing potential with no effective contraceptive method
14. Participant who participated in any drug clinical trial within the last 3 months prior to screening visit
15. History of severe hypersensitivity to rExenatide-4 or any product components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from Baseline to Week 30 | Baseline (Day 1) to Week 30
  Change in HbA1c from Baseline (Day 1) to study termination (Week 30)

SECONDARY OUTCOMES:
The number of subjects achieving HbA1c target values of < 7% and ≤ 6.5% by Week 30 | Baseline (Day 1) and Week 30
  The number of subjects achieving HbA1c target values of < 7% and ≤ 6.5% by study termination (Week 30)
Change in body weight from Baseline to each intermediate visit and Week 30 | Baseline (Day 1), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 30
  Change in body weight (kg) from Baseline to each intermediate visit and Week 30
Change in FPG from Baseline to each intermediate visit and Week 30 | Baseline (Day 1), Week 2, Week 4, Week, 6, Week 12, Week 18, Week 24, Week 30
  Change in Fasting Plasma Glucose from Baseline to each intermediate visit and Week 30
Change in 7-SMBG from Baseline to Week 16，Week 24 and Week 30 | Baseline, Week 16，Week 24 and Week 30
  Change in glucose measurements before and 2h after the start of the morning,midday,and evening meals, and at bedtime from Baseline to Week 16，Week 24 and Week 30

CONTACTS AND LOCATIONS:
Overall Officials: linong Ji, Ph.D, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No